CLINICAL TRIAL: NCT03523676
Title: Evaluation of Red Cell Distribution Width to Predict New-onset Atrial Fibrillation in Critically Ill Sepsis Patients
Brief Title: Use of Red Cell Distribution Width for Prediction of New-onset Atrial Fibrillation in Critically Ill Sepsis Patients
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed, Clinical researcher, Ain Shams University
Other Study IDs: R33 /2018
Record Dates: First submitted 2018-05-02; First posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Atrial Fibrillation New Onset
MeSH Terms: interventions — Erythrocyte Indices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: sepsis patients who did not develop atrial fibrillation during ICU stay
  Interventions: Diagnostic Test: Red Cell Distribution Width
- Group B: sepsis patients with newly developed atrial fibrillation during ICU stay
  Interventions: Diagnostic Test: Red Cell Distribution Width

INTERVENTIONS:
Diagnostic Test: Red Cell Distribution Width

SUMMARY:
Red cell distribution width variations are increased in a variety of medical conditions such as congestive heart failure, acute myocardial infarction, pulmonary embolism, pneumonia, critical illness, and cardiac arrest , and is a predictor of mortality in the general population..

DETAILED DESCRIPTION:
This study was done retrospectively on sepsis patients admitted to intensive care units. data will be retrieved from patient medical records. The primay end point will be occurrence of new-onset AF during ICU stay. The secondary outcomes will be 28-day mortality.

The presence of anisocytosis or RDW variations has been classicaly used as a test for iron deficiency anemia. Increasing evidence points to its potential as a predictor for various conditions such as heart failure , malignancy, ischemic heart disease and sepsis.

Study investigators will examine the relationship between RDW levels and incidence of atrial fibrillation in critically ill sepsis patients as well as 28-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* For all patients According to Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3) , adult patients with suspected infection are identified, having quickSOFA (qSOFA) score meeting ≥2 of the following criteria: respiratory rate of 22/min or greater, altered mentation, or systolic blood pressure of 100 mmHg or less
* Sepsis patients with newly developed Atrial fibrillation during ICU stay.

Exclusion Criteria:

All patients with concomitant valvular disease, cardiomyopathy, cardiac dysrhythmias, previous cardiac surgery, secondary hypertension, hyperthyroidism, severe head injury, stroke, coma, acute coronary artery disease or underlying cardiac dysfunction[cardiac index (CI) <2.2 l/min/m 2 ], severe liver disease (Child-Pugh grade C), chronic renal failure were excluded from the study. In addition, pregnant patients were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 patients of both sexes were enrolled in this study. They were admitted to the general ICU of Ain Shams University Hospitals with sepsis or septic shock
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-03-10 (Actual)

PRIMARY OUTCOMES:
New-Onset atrial fibrillation , confirmed by electrocardiographical assessment | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Diaaeldein Ibrahim, MD, Study Director — Ain Shams University

IPD SHARING:
Plan to Share IPD: Undecided